CLINICAL TRIAL: NCT05975619
Title: A Prospective Imaging Study of Target Definition and Radiation Planning Workflows on the Integrated TrueBeam-HyperSight System for Patients Receiving Radiation Therapy
Brief Title: A Prospective Imaging Study of the Integrated TrueBeam-HyperSight CBCT System
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Varian, a Siemens Healthineers Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VAR-2023-03
Record Dates: First submitted 2023-07-17; First posted 2023-08-04 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Head and Neck Cancer; Thoracic Cancer; Abdominal Cancer; Pelvic Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Pelvic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-arm, single-site feasibility study designed to generate data describing the quality and applicability of on-couch high-performance CBCT imaging technology.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- HyperSight Imaging arm (Experimental): Subjects are imaged with the new HyperSight CBCT imaging system.
  Interventions: Device: HyperSight imaging

INTERVENTIONS:
Device: HyperSight imaging — Subjects are scheduled for 1 to 5 HyperSight imaging sessions, which will occur on the same days as their standard clinical visits during planning and treatment delivery. A total of 5 to 10 HyperSight CBCT images will be acquired over all imaging sessions.

SUMMARY:
Cone beam computed tomography (CBCT) images are routinely used in radiation treatment delivery workflows to align patients with the treatment beam. Conventional CBCT image quality is sufficient for this task but not good enough for other radiotherapy-related tasks, such as contouring anatomical structures and calculating radiation dose distributions. HyperSight is a new CBCT imaging system manufactured by Varian Medical Systems. The purpose of this study is to evaluate the integration of the HyperSight imaging system with Varian's TrueBeam radiotherapy system, a linear accelerator with a C-arm gantry that rotates about the patient to delivery radiation to the target malignancy. HyperSight CBCT images will be acquired prospectively from patients who are receiving radiation treatment. The HyperSight/TrueBeam system will be used for imaging only; patients receive their radiation treatment on cleared devices and no aspect of their treatment is affected by participation in the study. HyperSight images collected during the study will be evaluated for quality and utility and compared to conventional CBCT images as well as fan beam CT images used for treatment planning.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is scheduled to receive radiation therapy to one of the following anatomical sites: head and neck/brain, thorax, abdomen, pelvis.
2. Patient is at least 18 years of age.
3. If the patient will be receiving IV contrast on study, patient must have adequate renal function as defined by an estimated glomerular filtration rate (eGFR) of >30.

   Note: if no IV contrast will be administered on study, patient may enroll without creatinine level documented. Contrast eligibility will be determined as per Appendix A.
4. If the patient is a woman of childbearing potential, patient must have a negative pregnancy test within 30 days of enrollment and prior to any study imaging. Contraceptive use is not an adequate documentation of no chance of pregnancy.

Exclusion Criteria:

1. Patient is unwilling or unable to sign an IRB-approved written informed consent document.
2. Patient is part of a vulnerable population (per ISO 14155:2020, "individuals who are unable to fully understand all aspects of the investigation that are relevant to the decision to participate, or who could be manipulated or unduly influenced as a result of a compromised position, expectation of benefits or fear of retaliatory response").

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-29 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Feasibility of using HyperSight CBCT images for radiation treatment planning. | 1-9 weeks
  The percentage of images that are of sufficient quality for patient treatment plan generation.

OTHER OUTCOMES:
OAR delineation | 1-9 weeks
  Comparison of organ at risk (OAR) delineation on TrueBeam-HyperSight CBCT images to OAR delineation on conventional CBCT images, as well as on fan beam CT.
Image quality - quantitative | 1-9 weeks
  Assessed through calculated image metrics.
Image quality - qualitative | 1-9 weeks
  Assessed through expert observer evaluations of the images for utility in the radiotherapy workflow.
Patient anxiety | 1-9 weeks
  Assessed through a patient survey using the validated Six-Item State Anxiety Scale derived from the State-Trait Anxiety Inventory. Each of the six items in the survey are assigned a score from 1 to 4 indicating the patient's agreement to a statement such as "I am tense", where 1 represents "Not at all", and 4 represents "Very much so".
Treatment plan quality | 1-9 weeks
  Assessed through comparison of dose-volume histogram (DVH) metrics extracted from the re-calculation of the patient's treatment plan on the HyperSight CBCT to DVH metrics from the patient's treatment plan originally calculated on the pre-treatment simulation fan-beam CT.
Patient clearance | 1-9 weeks
  Evaluated by the number of instances where patient positioning and/or custom immobilization devices created for their standard-of-care radiation therapy were incompatible with system geometries of the TrueBeam-HyperSight system during imaging and clearance checks.
Timing of image registration | 1-9 weeks
  The time required to register a HyperSight CBCT to the patient's reference CT simulation image.
Confidence in image registration | 1-9 weeks
  Assessed through a user-rated confidence (measured using a three-point scale: low/moderate/high).
Impact of off-axis imaging on Hounsfield Unit accuracy | 1-9 weeks
  In images where the center of rotation is shifted, the impact of the off-axis imaging on the HU accuracy will be evaluated by comparing dose-volume histogram metrics between the treatment plan generated on the off-axis HyperSight CBCT and DVH metrics from the patient's treatment plan, calculated on a fan-beam CT that does not have the same limited field of view as the CBCT.
Impact of image acquisition time on clinical efficiency | 1-9 weeks
  Timing of workflow steps and processes including setup, imaging, alignment, and door-to-door time as compared to standard-of-care imaging processes, and compared to clinical models for hypothetical, generic clinics, using a time-driven, activity-based cost model.
Feasibility of obtaining respiratory gated HyperSight CBCT | 1-9 weeks
  Assessed through evaluation of internal motion volumes of organs-at-risk and targets, relative to diaphragm and/or vertebral body position, as compared to 4D-CT from standard-of-care simulation imaging.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No